CLINICAL TRIAL: NCT00371722
Title: A Randomized Controlled Trial Evaluating Appendectomy at the Time of Cesarean Section
Brief Title: Appendectomy Versus no Appendectomy With Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Obstetrical Consultants (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 02-052
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Cesarean Delivery; Appendectomy
Keywords: Cesarean section; Appendectomy
MeSH Terms: interventions — Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Appendectomy

SUMMARY:
Women having cesarean section will be divided into two groups - cesarean section alone or cesarean section with appendectomy. The purpose is to see if the appendectomy can be done without adding any complications to the maternal post-operative course. The hypothesis is that there is no increased incidence of wound infection, post-operative morbidity or longer hospital stay associated with elective appendectomy at the time of Cesarean Section.

DETAILED DESCRIPTION:
Even though the incidence of appendicitis has decreased significantly since the advent of antibiotics, the disease process is still quite ubiquitous in many patient populations. The incidence of appendicitis in women over 20 and under 50 years of age is significant. The annual incidence of appendicitis in women aged 17 to 64 years of age is 1.9 per 1000. In the population aged 15 to 19 years of age, the risk of developing appendicitis is 1 in 99 in each year of this 4-year period. Diagnosing appendicitis in pregnancy poses a great challenge for the obstetrician because the appendix is displaced during pregnancy, nausea is common in pregnancy, direct abdominal signs are variable as well. The incidence of proven appendicitis approximates 1 in 1500 deliveries. Maternal and fetal mortality and morbidity are increased when appendicitis is associated with pregnancy, and the risks rise significantly if perforation and peritonitis occur. Fetal loss, which is between 10 and 20% in most reports, is mainly due to preterm labor or intrauterine death, particularly when perforation occurs. There are three main reasons to perform an incidental appendectomy (at the time of cesarean section): To reduce future mortality and morbidity from appendicitis in women of childbearing age; to eliminate undiagnosed incidental pathology in the appendix; and to eliminate the appendix from diagnostic consideration when the patient presents with abdominal or pelvic complaints. There will be 100 subjects taking part in the study. Standard post operative care will be administered with the only difference in the two groups being the operative procedure (appendectomy or no appendectomy).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years age
* No previous appendectomy
* Adequate pain control for cesarean section
* Able to give informed consent

Exclusion Criteria:

* Previous appendectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2002-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Post-operative wound infection

SECONDARY OUTCOMES:
Post-operative fever
Post-operative length of hospital stay
Post-operative need for pain control

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Adair, MD, Principal Investigator — Regional Obstetrical Consultants; UT Chattanooga OB-GYN Department
Locations (1):
- Erlanger Medical Center, Chattanooga, Tennessee, United States